CLINICAL TRIAL: NCT01433601
Title: A Randomised Controlled Trial to Assess Antiretroviral Treatment Strategies in Relation to Adherence, Resistance and Virological Treatment Failure
Brief Title: Antiretroviral Treatment Strategies in Relation to Adherence, Resistance and Virological Treatment Failure
Acronym: DotArv
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Mattias Larsson, MD PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DotArv_Vietnam
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Adherence; Peer support; Treatment failure
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self Supervised Treatment (SST) (No Intervention): Treatment according to the National Treatment Guidelines in Vietnam including treatment counseling before initiation of ART and clinical follow up every 3 months. The patient is self responsible to take the drugs and no additional adherence support is provided.
- Enhanced Treatment Support (ETS) (Experimental): Treatment according to the National Treatment Guidelines in Vietnam including treatment counseling before initiation of ART and clinical follow up every 3 months. In addition adherence support is provided according to the description under intervention.
  Interventions: Behavioral: Enhanced Treatment Support (ETS)

INTERVENTIONS:
Behavioral: Enhanced Treatment Support (ETS) — An "internal supporter" - family member or other person trusted by the patient is trained to fill in a checklist whether the drugs has been taken and if this was observed. An"external supporter" - a peer selected PLWHA visit the patient twice weekly the first two months. The external supporter follows a checklist and ask about general well being, psychological problems or adverse drugs reactions as well as go through the adherence since last visit, using the internal supporter checklist. If the adherence is good, the number of visits are decreased to once weekly after two months, if not, the number of visits are intensified. If there are any symptoms of opportunistic infections, immunological reconstruction syndrome or adverse drug reactions the patient are refered for medical checkup.
  Other Names: Peer support; Directly Observed Treatment (DOT); Adherence support; Adherence counselling
  Arms: Enhanced Treatment Support (ETS)

SUMMARY:
This project aims to assess different antiretroviral treatment strategies, optimally controlled and conventional, in relation to drug resistance and virological treatment failure. A Randomised Controlled trial (RCT) where Vietnamese HIV+ patients with CD4+ T-cells <200/ul are randomized into either enhanced treatment support (ETS) through peer supporters or The National AIDS Control Program recommended self supervised treatment (SST). The treatment strategies will be assessed and compared in relation to treatment adherence and drug resistance development with virological treatment failure as primary endpoint. The results from this project will lead to an increased knowledge in relation the impact of treatment support on adherence, virological suppression and resistance development and have an impact on HIV treatment policies in low income settings globally.

DETAILED DESCRIPTION:
Aim To study the impact of patient support on selective drug pressure, defined by semi-quantitative assessments of adherence, on the viral suppression and resistance development through a randomised controlled trial of HIV positive patients randomised in enhanced treatment support (ETS) and self supervised treatment (SST).

Specific Objectives

1. To create a study population 600 HIV+ patients with CD4+ T-cell count of <200/ul and randomize in two different treatment cohorts, enhanced treatment support (ETS) and conventional self-supervised treatment (SST).
2. To monitor the patients using semi-quantitative assessments of adherence, clinical status including clinical examinations (every 3 months), viral load and CD4+ T-cell count (every 6 months) during 24 months with virological treatment failure as primary endpoint.
3. To compare the ETS and SST cohorts with respect to the primary endpoint, virological treatment failure, in relation to the semi-quantitative assessments of adherence and to analyse the mechanism of selective drug pressure for the development of resistance including resistance in minor viral subpopulations.
4. To conduct a cost effectiveness assessment comparing ETS and SST with respect to the labour and infrastructural cost, virological treatment failure and change to second line therapy.

The study is conducted in Quang Ninh Province, the area hardest hit by the HIV epidemic in Vietnam with a known HIV+ prevalence above 1%. A study population of 600 HIV+ patients with CD4+ T-cell count of <200 are being be recruited in four districts, Ha Long, Uong Bi, Yen Huong and Dong Trieu. Each HIV+ person is examined according to WHO guidelines. HIV+ persons receive a complete physical examination, clinical staging of HIV infection, opportunistic infections including HBV, HCV and tuberculosis. Laboratory testing will include Full blood count, CD4+ T-cell count, viral load using the affordable and simple ELISA based ExaVirR viral load test (http://www.cavidi.se), liver enzymes, PAP smear and pregnancy test for women. If indicated (e.g. prolonged cough) chest X-ray, sputum microscopy for AFB are done.

Opportunistic infections in HIV+ patients are treated according to national guidelines. HIV+ persons receive counselling including information about the disease and the plan for care and treatment, follow-up visits, nutrition and living, prevention of HIV transmission including safe sex, harm reduction measures, the use of birth control methods and prevention of mother to child HIV transmission.

Inclusion and exclusion criteria's are described below. The patients will be randomised into two equally large cohorts, receiving either of two different treatment strategies a) enhanced treatment support (ETS) (described below) and Self-supervised treatment (SST). Co-infections are assessed, diagnosed and the treatment adjusted according to the national guidelines for such situations. The patients are studied with respect to: (i) virological treatment failure, (ii) adverse effects. (iii) patient's adherence to treatment strategy. First drug regimen for all patients including stavudine, lamivudine, nevirapine or efavirenz dosages, follow up for adverse effects and regimen alteration are done according to national guidelines. The health care workers are trained in regular monitoring of patients and implementation of optimal treatment strategy. All procedures and treatment will follow the national guidelines. Follow up consultations including physical examinations and tests are done every 3 month.

The tests will include full blood count, CRP, electrolytes, liver enzymes as well as other indicated. Viral load are monitored every 6 month and CD4+ T-cell count every 12 month.

The number of patients needed for each arm of the experiment was estimated assuming a difference between arms of 15 percent units for treatment failure and corresponding baseline percentage of 20%. Requiring a power of 80% and a significance level of 5% the necessary number is about 300 per arm. Inflating the size by 30% to compensate for expected loss to follow up the investigators get just under 300 patients per arm. The assumptions about differences are based on the following: a) Differences larger than 10% units in virological treatment failure are indications for review and modification of treatment strategies; b) group differences in virological treatment failure less the 20% are unlikely to lead to policy changes in Vietnam. The discussion above uses a binary variable like failure/no failure. Performing analysis on quantitative variables like CD4 T-cell readings, which are more informative, will in some cases have considerably higher power than the corresponding binary.

In the ETS strategy an "internal supporter", family member or other person trusted by the patient, is trained to fill in a checklist whether the drugs has been taken and if this was observed. An"external supporter" - a peer selected PLWHA visit the patient twice weekly the first two months. The external supporter follows a checklist and ask about general well being, psychological problems or adverse drugs reactions as well as go through the adherence since last visit, using the internal supporter checklist. If the adherence is good, the number of visits are decreased to once weekly after two months, if not, the number of visits are intensified. If there are any symptoms of opportunistic infections, immunological reconstruction syndrome or adverse drug reactions the patient are refered for medical checkup.. In SST the patient will self be responsible to take the drugs. At initiation treatment counseling are provided. In both groups the drugs are provided in a pre-packed dosage form for easy remembering and counting of the pills.

The patients are followed for 24 months and monitored through clinical examination (each 3 months), viral load in plasma (each six months), CD4- T-cell counts (each 6 months) and assessment of well-being (every 3 months). Adherence among patients are assessed using Contextualised Adult AIDS Clinical Trials Group (AACTG) Adherence Instruments (Chesney et al, 2000). AACTG Adherence Instruments consists of two questionnaires and the first questionnaire is specifically developed to be used for baseline assessment of adherence. The second questionnaire version is developed for assessment of adherence during follow-up visits. Adherence are assessed using the AACTG Adherence Instruments every third month in both the ETS and SST groups. One person is present at the clinic to answer questions regarding the questionnaire and provide help if necessary. Adherence is also measured by pill count conducted by the External supporters, enabling calculation of the proportion of drugs remaining out of the total amount of prescribed drugs. Assessment of side effects according to WHO suggested monitoring and management of ARV drugs are done together with the clinical examination each three months.

The primary endpoint is virological treatment failure defined as a viral load of 1 fg reverse transcriptase activity/ml, corresponding to 200 copies/ml, at 1 year and 2 years after starting treatment. Drug Resistance is determined using a selective real-time PCR for the detection of the critical mutations in the RT-gene, as a marker for whether virological treatment failure that occurs with wild-type virus or resistant virus. The secondary endpoints immunological treatment failure (no rise in CD4+ T-cell count at 1 year) and clinical treatment failure as defined by a new AIDS defining illness or death due to HIV/AIDS (including TB and opportunistic infection) after starting treatment.

Costing of the two different strategies will be carried out by collecting monetary data of expenses of drugs, test, allowance and other expenses from perspective of the HIV/AIDS treatment provider during ART. The investigators follow the basic principles of activity-based costing by identifying all activities necessary to provide the EST and SST and then calculate the costs of carrying out each activity. Costs for each activity comprise recurrent and capital costs, direct and indirect costs. Recurrent costs are the routine costs of resources that are consumed within a year, i.e., non-capital items such as labor and medical supplies. Capital costs represent the annual portion of the cost of durable HIV Sida DOTARV assets. Effectiveness will be measured by percentages of patients with virological treatment failure defined as Viral Load>400 copies/ml.

The statistical analysis mainly consists in the comparison between the two groups with respect to the defined primary endpoint, virological treatment failure, and possibly the secondary endpoints immunological treatment failure and clinical treatment failure, in relation to the semi-quantitative assessments of adherence. Basically standard statistical methods will be used. Regression models with outcome as the dependent variable and a group indicator together with person characteristics as independent variables will be the main approach. For binary outcomes, logistic regression will be used. Attention has to be paid to the particular, often skewed, distributions of variables like CD4+ T-cell counts and viral load. Transformations or the use of non-parametric approaches are likely to be necessary if such measures are not dichotomised and used in linear regression. The correlation between drug resistance to the used drugs (stavudine, lamivudine, nevirapine) and adherence will be statistically analysed in order to study whether the basic mechanisms of selective drug pressure result in a concave or bell-shaped resistance - adherence relationship, for these drugs during ETS or SST in a low-income setting.

The investigators will strictly comply with widely recognized international texts and codes of practice including the Helsinki agreement. In this project one patient cohort will receive ETS and the other SST. Both the OTC and SST cohorts will be encouraged to proceed regularly with their drug treatment and to present difficulties that they may encounter in doing so. For the project period, the project will meet the costs of ARV for the cohorts. Patients' biological samples are collected and used only after written consent. All specimens are coded to protect the identity of patients and to ensure confidentiality. Patients are recruited in a consecutive manner without regard to race or other exclusion considerations. Confidentiality is assured by using codes for patient identification, and confidentially laws will be strictly observed when processing human clinical information. No patient identifying information will be published or available after the requisite clinical data have been collected, and consent will be obtained for the use of all data and tissues. Data is accessible only to members and coordinators of the tissue procurement facility and research team, under approved guidelines.

ELIGIBILITY:
Inclusion Criteria:

* WHO stage IV of HIV disease, regardless of the CD4 count
* WHO stage III of HIV disease with a CD4 count < 350/mm3
* WHO stages I or II with a CD4 count < 200/mm3

Exclusion Criteria:

* Pregnancy
* Ongoing severe opportunistic infections
* Institutionalized patients.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 640 (Actual)
Dates: Start 2007-08; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Virological treatment failure | 24 months
  HIV viral load of 1 fg reverse transcriptase activity/ml, corresponding to 200 copies/ml, at 1 year and 2 years after starting treatment.

SECONDARY OUTCOMES:
Immunological treatment failure | 24 months
  Immunological treatment failure
  * CD4 count returns to or falls below pre-therapy baseline level or
  * 50% decline from the on-treatment peak value since the initiation of ART (if known); or
  * CD4 count < 100 cells/mm3 after a year without any increase.
Clinical treatment failure | 24 months
  Occurrence or recurrence of stage 4 diseases or conditions after at least 6 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Larssson, Md PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Hanoi Medical University, Hanoi, Hanoi, Vietnam

REFERENCES:
- [Derived] Cuong DD, Sonnerborg A, Van Tam V, El-Khatib Z, Santacatterina M, Marrone G, Chuc NT, Diwan V, Thorson A, Le NK, An PN, Larsson M. Impact of peer support on virologic failure in HIV-infected patients on antiretroviral therapy - a cluster randomized controlled trial in Vietnam. BMC Infect Dis. 2016 Dec 16;16(1):759. doi: 10.1186/s12879-016-2017-x. PMID 27986077
- [Derived] Van Tam V, Cuong DD, Alfven T, Phuc HD, Chuc NT, Hoa NP, Diwan V, Larsson M. HIV sero-discordance among married HIV patients initiating anti-retroviral therapy in northern Vietnam. AIDS Res Ther. 2016 Nov 15;13:39. doi: 10.1186/s12981-016-0124-9. eCollection 2016. PMID 27891160
- [Derived] Cuong do D, Thorson A, Sonnerborg A, Hoa NP, Chuc NT, Phuc HD, Larsson M. Survival and causes of death among HIV-infected patients starting antiretroviral therapy in north-eastern Vietnam. Scand J Infect Dis. 2012 Mar;44(3):201-8. doi: 10.3109/00365548.2011.631937. Epub 2011 Nov 28. PMID 22122590